CLINICAL TRIAL: NCT07354074
Title: A Phase II, Multicenter, Open-label, Single Arm Study to Evaluate the Safety and Efficacy of Asciminib in Pediatric Participants Newly Diagnosed or Previously Treated With Philadelphia Positive Chronic Myelogenous Leukemia in Chronic Phase (Ph+ CML-CP) With or Without Known T315I Mutation
Brief Title: Study to Determine the Efficacy and Safety of Asciminib in Pediatric Patients With Ph+ CML-CP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001I12202; 2025-522138-29 (Registry Identifier: EU CTIS)
Expanded Access: NCT04360005 (Available)
Record Dates: First submitted 2026-01-15; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelogenous Leukemia; Leukemia, Myelogenous, Chronic, Philadelphia Chromosome Positive
Keywords: Asciminib; ABL001; Pediatric participants; Philadelphia chromosome positive chronic myeloid leukemia in chronic phase; Ph+ CML-CP; tyrosine kinase inhibitor; TKI; Molecular Response; MR; CML; Chronic phase; T3151; Ph+
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — asciminib

STUDY DESIGN:
Intervention Model Description: Three cohorts of Ph+ CML-CP pediatric participants receive asciminib: (1) newly-diagnosed without known T315I mutation; (2) resistant or intolerant to previous TKI without known T315I mutation; and (3)with known T315I mutation irrespective of prior TKI treatment. Outcomes are evaluated separately for each cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): This study will enroll pediatric patients (≥ 1 and < 18 years of age) with newly diagnosed or previously treated with Philadelphia positive Chronic Myelogenous Leukemia in Chronic Phase (Ph+ CML-CP) with or without known T315I mutation
  Interventions: Drug: Asciminib single agent

INTERVENTIONS:
Drug: Asciminib single agent — Asciminib (labelled as ABL001) administered as 40 mg tablet (adult formulation) or as 1 mg film-coated granules mini-tablets (pediatric formulation)
  Other Names: ABL001

SUMMARY:
The aim of this study is to support development of asciminib in the pediatric population (1 to < 18 years) with Ph+ CML-CP. The study will evaluate the efficacy and safety of asciminib in pediatric formulation (weigh-based dose, fed state) or adult formulation (fasted) in newly diagnosed and resistant or intolerant Ph+ CML-CP with or without T315I mutation.

DETAILED DESCRIPTION:
This is a multi-center, open-label, single arm study of asciminib in pediatric participants aged

1 to <18 years old with Ph+ CML-CP newly diagnosed and previously treated with TKI treatment, with or without T315I mutation.

The study population will consist of three cohorts of Ph+ CML-CP pediatric participants:

* Newly-diagnosed Ph+ CML-CP participants without known T315I mutation
* Ph+ CML-CP participants resistant or intolerant to previous TKI without known T315I mutation
* Ph+ CML-CP participants with known T315I mutation irrespective of prior TKI treatment

There is no fixed duration of study treatment for the participants. The study will end 5 years (240 weeks) after the last enrolled participants received their first dose of treatment in the study. The objective is to have enough follow up for safety, including growth and development and efficacy.

ELIGIBILITY:
Key Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Male or female participants 1 and < 18 years of age at study enrollment
3. Diagnosis of CML-CP (Apperley et al 2025) with cytogenetic confirmation of Philadelphia positive (Ph+) chromosome
4. For participants with CML-CP newly diagnosed within 3 months of screening OR 5 For participants with CML - CP with high risk of developing resistance or intolerance to previous TKI:

   1. Unfavourable response to TKI is defined following the Apperley et al 2025 guidelines as:

      * At three months after the initiation of therapy: BCR::ABL1 ratio > 10% IS (if confirmed within 1-3 months)
      * At six months after the initiation of therapy: BCR::ABL1 ratio > 10% IS
      * At twelve months after initiation of therapy: BCR::ABL1 ratio > 1% IS
      * At any time loss of previous response
      * At any time emergent resistant BCR::ABL1 mutations or high-risk ACA from prior TKI treatment as per local test results
   2. Intolerance to TKI is defined as:

      * Non-hematologic intolerance: participants with grade 3 or 4 toxicity while on therapy (in which case the patient is eligible whether or not there was a dose reduction); or with persistent grade 2 toxicity unresponsive to optimal management including dose adjustments (unless dose reduction is not considered in the best interest of the patient if response is already suboptimal)
      * Hematologic intolerance: participants with grade 3 or 4 toxicity (absolute neutrophil count [ANC] or platelets) while on therapy that is recurrent after dose reduction to the lowest doses of the TKI

6. Evidence of typical BCR::ABL1 transcript [e14a2 and/or e13a2] at the time of screening which are amenable to standardized RQ-PCR quantification.

7. Performance status: Karnofsky ≥ 50% for participants ≥ 16 years of age, and Lansky ≥ 50 for participants < 16 years of age at the time of screening.

Key Exclusion Criteria:

1. Known second chronic phase (CP) of CML after previous progression to Accelerated Phase (AP)/Blast Phase (BP).
2. Previous treatment with a hematopoietic stem-cell transplantation.
3. Patient planned to undergo allogeneic hematopoietic stem cell transplantation
4. Known presence of a BCR::ABL1 mutation with known resistance to study treatment in accordance with the most recent public version of international CML clinical guidelines (e.g. NCCN CML treatment guidelines v 1.2026 and Apperley et al 2025) any time prior to study entry

Other inclusion/exclusion criteria may apply.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-06-04 (Estimated); Primary Completion 2033-02-23 (Estimated); Study Completion 2033-02-23 (Estimated)

PRIMARY OUTCOMES:
MMR at Week 48 | 48 weeks
  MMR is defined as BCR::ABL1 IS ≤0.1%. MMR is defined as a ≥ 3.0 log reduction in BCR::ABL1 transcripts compared to the standardized baseline equivalent to ≤ 0.1 % BCR::ABL1/ABL % by international scale as measured by RQ-PCR.

SECONDARY OUTCOMES:
MMR at Week 96 | 96 weeks
  MMR is defined as BCR::ABL1 IS ≤0.1%. MMR is defined as a ≥ 3.0 log reduction in BCR::ABL1 transcripts compared to the standardized baseline equivalent to ≤ 0.1 % BCR::ABL1/ABL % by international scale as measured by RQ-PCR.
MMR at and by scheduled timepoints | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96
  MMR is defined as BCR::ABL1 IS ≤0.1%. MMR is defined as a ≥ 3.0 log reduction in BCR::ABL1 transcripts compared to the standardized baseline equivalent to ≤ 0.1 % BCR::ABL1/ABL % by international scale as measured by RQ-PCR.
Hematologic response at and by scheduled timepoints | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96
  Complete hematologic response (CHR) is defined as all of the following present for ≥ 4 weeks (which means present at least at 2 visits 4-week apart, with no intermediate visit showing no CHR):
  * White blood cell(s) (WBC) count < 10 x 10^9/L
  * Platelet count < 450 x 10^9/L
  * Basophils < 5%
  * No blasts and promyelocytes in peripheral blood
  * Myelocytes + metamyelocytes < 5% in peripheral blood
  * No evidence of extramedullary disease, including spleen and liver
Cytogenetic response at and by scheduled timepoints | 5 years
  Cytogenetic response is defined as follows:
  * Complete (CCyR) - 0% Ph+ metaphases
  * Partial (PCyR) - >0 to 35% Ph+ metaphases
  * Major* (MCyR) - 0 to 35% Ph+ metaphases
  * Minor (mCyR) - >35 to 65% Ph+ metaphases
  * Minimal - >65 to 95% Ph+ metaphases
  * None - >95 to 100% Ph+ metaphases Bone marrow aspirate for cytogenetic analyses will be performed at screening, and upon unfavorable response to treatment at the physician's discretion.
Time to response | 240 weeks after the last participant enrolled in the study received the first dose of treatment
  Time to the first response is defined as: date of the first documented occurrence of the response or time from first study drug intake to first response - date of the first study treatment intake + 1.
Duration of response (limited to the binary response endpoints) | 240 weeks after the last participant enrolled in the study received the first dose of treatment
  Duration of response is defined as the time between the date of the first documented occurrence of the response and the earliest date of confirmed loss of the response, progression to accelerated phase/blast crisis (AP/BC) or CML-related death for participants in the respective Responder Set.
Time to treatment failure (TTF) | 240 weeks after the last participant enrolled in the study received the first dose of treatment
  TTF is defined as the time from the first study drug intake to the first/earliest documented date of any of the following events: unfavorable response to treatment, confirmed loss of MMR at any time while on study treatment and discontinuation from study treatment due to any reason.
Time to disease progression | 5 years
Event-free survival (EFS) | 240 weeks after the last participant enrolled in the study received the first dose of treatment
  EFS is defined as the time from the first study drug intake to the earliest occurrence of the following events: unfavorable response to treatment, confirmed loss of MMR at any time while on study treatment, discontinuation from the study treatment due to an adverse event (AE) and death due to any cause.
Overall survival (OS) | 240 weeks after the last participant enrolled in the study received the first dose of treatment
  OS is defined as the time from the first study drug intake to the date of death from any cause during the study (including death observed during the survival follow-up period after discontinuation of study treatment).
Growth: Height/length, weight, bone age measured by X-Ray | 240 weeks after the last participant enrolled in the study received the first dose of treatment
  To assess growth and sexual maturation. An X-ray of the left hand and wrist to assess bone age will be performed at screening and every 48 weeks until end of treatment (EOT). This assessment will no longer be required for participants once bone maturity in post-puberty stage is confirmed by the last X-ray.
Sexual maturation: Height/length, weight, bone age measured by Tanner staging | 240 weeks after the last participant enrolled in the study received the first dose of treatment
  To assess growth and sexual maturation. Tanner staging will be based on external genitalia, breast and pubic hair examination. Tanner staging will be assessed for all study participants at screening. Participants who do not have a baseline Tanner Stage of 5 will continue to be assessed every 24 weeks until achievement of Tanner Stage 5 on both secondary sexual characteristics or EOT, whichever comes first. Once a participant reaches stage 5, examinations do not need to be conducted anymore. For all male participants, Tanner Stage 5 will be achieved once the participant has demonstrated both stage 5 genitalia development and stage 5 pubic hair development. For all female participants, Tanner Stage 5 will be achieved once the participant has demonstrated both stage 5 breast development and stage 5 pubic hair development.
PK parameters of asciminib: AUClast | Week 2, Day 1 at 1, 3 and 6 hours post dose
  AUClast: The AUC from time zero to the last measurable concentration sampling time.
PK parameters of asciminib: AUCtau | Week 2, Day 1: pre dose (0 hour), Week 2: Day 1 at 1, 2, 3, and 6 hours post-dose
  AUCtau: The AUC calculated to the end of a dosing interval (tau) at steady-state.
PK parameter of asciminib: Cmax | Week 2, Day 1 at 1, 3, and 6 hours post dose
  Cmax is the maximum (peak) observed plasma drug concentration after single dose administration.
PK parameter of asciminib: Tmax | Week 2, Day 1 at 1, 3, and 6 hours post dose
  Tmax is the time to reach maximum (peak) plasma drug concentration (h) after administration.
PK parameter of asciminib: Ctrough | Week 2, Day 1: pre-dose (0 hr), Week 24: pre-dose (0 hr), Week 48: Pre-dose (0 hr)
  Ctrough refers to the lowest concentration a drug reaches in the bloodstream immediately before the next dose is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com